CLINICAL TRIAL: NCT02069015
Title: Achieving Blood Pressure Control Through Enhanced Discharge
Acronym: AchieveBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Julie Gleason-Comstock, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BCBSMF 1956.11
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
Keywords: Patient education; Hypertension; Patient activation
MeSH Terms: conditions — Hypertension; Patient Participation | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced discharge (Experimental): Patient education about hypertension delivered through a touch-screen kiosk at 4 time points in addition to standard discharge.
  Interventions: Behavioral: Patient education
- Standard discharge (No Intervention): Standard discharge is patient instruction, instructions for follow-up to primary care and medication/prescription

INTERVENTIONS:
Behavioral: Patient education — Patient education on hypertension delivered through a touchscreen kiosk.
  Arms: Enhanced discharge

SUMMARY:
The primary aim of the study is to determine if enhanced discharge from the emergency department will improve blood pressure control and self-care management. Enhanced discharge will include a hypertension intervention delivered by a touch-screen kiosk over a three month period.

DETAILED DESCRIPTION:
A targeted sample of patients with uncontrolled blood pressure at the time of their emergency department visit discharge will be randomized into either standard or enhanced discharge. To control for medication effects in achieving blood pressure control, both groups will receive similar blood pressure medication while actively participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Present with uncontrolled blood pressure to the emergency department (>140/90 for non-diabetics and >130/80 for diabetics)
* Self-reported history of hypertension

Exclusion Criteria:

* End-stage renal disease
* No history of hypertension
* Do not present with uncontrolled blood pressure

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Gleason-Comstock, PhD, Principal Investigator — Wayne State University; Phillip D Levy, MD, Principal Investigator — Wayne State University
Locations (1):
- Detroit Receiving Hospital Emergency Department, Detroit, Michigan, United States

REFERENCES:
- [Background] Gleason-Comstock JA, Streater A, Jen KL, Artinian NT, Timmins J, Baker S, Joshua B, Paranjpe A. Consumer health information technology in an adult public health primary care clinic: a heart health education feasibility study. Patient Educ Couns. 2013 Dec;93(3):464-71. doi: 10.1016/j.pec.2013.07.010. Epub 2013 Aug 12. PMID 23948646
- [Background] Levy PD, Cline D. Asymptomatic hypertension in the emergency department: a matter of critical public health importance. Acad Emerg Med. 2009 Nov;16(11):1251-7. doi: 10.1111/j.1553-2712.2009.00512.x. Epub 2009 Oct 20. PMID 19845553
- [Background] Levy P, Ye H, Compton S, Zalenski R, Byrnes T, Flack JM, Welch R. Subclinical hypertensive heart disease in black patients with elevated blood pressure in an inner-city emergency department. Ann Emerg Med. 2012 Oct;60(4):467-74.e1. doi: 10.1016/j.annemergmed.2012.03.030. Epub 2012 May 31. PMID 22658278
- [Background] Gleason-Comstock J, Streater A, Ager J, Goodman A, Brody A, Kivell L, Paranjpe A, Vickers J, Mango L, Dawood R, Levy P. Patient education and follow-up as an intervention for hypertensive patients discharged from an emergency department: a randomized control trial study protocol. BMC Emerg Med. 2015 Dec 21;15:38. doi: 10.1186/s12873-015-0052-3. PMID 26691646
- [Background] Gleason-Comstock J, Streater A, Goodman A, Janisse J, Brody A, Mango L, Dawood R, Levy P. Willingness to pay and willingness to accept in a patient-centered blood pressure control study. BMC Health Serv Res. 2017 Aug 7;17(1):538. doi: 10.1186/s12913-017-2451-5. PMID 28784120
- [Result] Gleason Comstock J, Janisse J, Streater A, Brody A, Goodman A, Zhang L, Mango L, Dawood R, Costello W, Patton S, Paranjpe A, Welsh C, Welch R, Levy P. Efficacy of enhanced emergency department discharge for chronic hypertension management - Results of a randomized controlled trial. Contemp Clin Trials Commun. 2020 Jul 18;19:100613. doi: 10.1016/j.conctc.2020.100613. eCollection 2020 Sep. PMID 32743119

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced Discharge | Standard Discharge
Started | 71 (Baseline and enrollment at Emergency Department (ED)) | 68
7 Day | 44 (7 day post ED discharge at Clinical Research Center (CRC)) | 45 (7 day post ED discharge at CRC)
30 Day | 38 (30 day post-discharge at CRC) | 43 (30 day post-discharge at CRC)
90 Day | 32 (90 day post ED discharge at CRC) | 35 (90 day post ED discharge)
Completed (Follow-up: 180 day post ED discharge) | 31 (180 post ED discharge at CRC) | 35 (180 day post ED discharge at CRC)
Not Completed | 40 | 33
Not completed — Lost to Follow-up | 39 | 32
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Patient education about hypertension delivered through a touch-screen kiosk at 4 time points in addition to standard discharge. Patient education on hypertension delivered through a touchscreen kiosk.
- Control: Standard discharge is patient instruction, instructions for follow-up to primary care and medication/prescription.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 71 | 68 | 139
Age, Categorical [Count of Participants; unit: Participants] — Post-discharge
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 69 | 67 | 136
    >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 38 | 68
  Male | 41 | 30 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 71 | 68 | 139
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Demographics [Count of Participants; unit: Participants]
  Education : <=HS/GED | 62 | 47 | 109
  Education : >=Associate Degree | 9 | 21 | 30
  Smoking Behavior : Never Smoked | 24 | 27 | 51
  Smoking Behavior : Ever Smoked | 47 | 41 | 88
  Diabetic Diagnosis : No Diabetic | 62 | 56 | 118
  Diabetic Diagnosis : Diabetic | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure (Systolic) at 180 Days
Description: Systolic Blood Pressure (SDB) at 180 days post-discharge
Time Frame: 180 days
Population: All participants for whom SBP were recorded at 180 days
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Control Group: All participants received hypertensive regimen
- Intervention Group: All participants received hypertensive regimen and education intervention
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 35 | 31
mmHg | 131 (18.0) | 131 (19.0)
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority; p < 0.001, paired t-test; Mean Difference = 0.05, 95% CI 2-sided [-4.781 to 6.906]

2. Secondary Outcome: Patient Activation Measure (PAM)
Description: Measure of how actively involved patient is in their medical care.
Time Frame: Baseline
Population: Patients discharged from the ED with uncontrolled hypertension assessed for PAM.
Measure: Count of Participants; unit: Participants
Groups:
- Patient Activation Measure (PAM): PAM sample at baseline is 4 levels; (1) awareness; (2) confidence; (3) action; (4) maintenance.
Arm/Group | Patient Activation Measure (PAM)
Number analyzed (Participants) | 128
Participants
  Control: number analyzed (Participants) | 63
  Control: Level 1 | 3
  Control: Level 2 | 19
  Control: Level 3 | 34
  Control: Level 4 | 7
  Intervention: number analyzed (Participants) | 65
  Intervention: Level 1 | 7
  Intervention: Level 2 | 20
  Intervention: Level 3 | 27
  Intervention: Level 4 | 11
  Total: Level 1 | 10
  Total: Level 2 | 39
  Total: Level 3 | 61
  Total: Level 4 | 18

3. Other Pre Specified Outcome: Emergency Department Visitation Rate
Description: Emergency department visits related to hypertension
Time Frame: Baseline to 180 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Cost Effectiveness
Time Frame: 180 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to 180 days
Arm/Group | Enhanced Discharge | Standard Discharge
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/68
Other Adverse Events (participants affected / at risk) | 0/71 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No